CLINICAL TRIAL: NCT06883721
Title: The Impact of Pilates Exercises on Pain, Posture, Range of Motion, Quality of Life, and Body Composition in Participants With Forward Head Posture: A Randomized Controlled Trial
Brief Title: Pilates Effects on Forward Head Posture: A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, yusuf yaşasın, Specialist Physiotherapist, PhD Student, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-02/02
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Pilates; Craniovertebral angle; Cervical stabilization; Randomized controlled trial; Neck pain; Posture; Rehabilitation
MeSH Terms: conditions — Neck Pain | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an experimental group (Pilates exercise group, n=18) or a control group (cervical stabilization exercise group, n=18) for an 8-week intervention period.
Who Masked: Outcomes Assessor
Masking Description: A blinded assessor performed all outcome measurements (NYPRS, VAS, goniometry, SF-36, anthropometric measurements).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilates Exercise Group (Experimental): Participants in this group performed Pilates exercises twice a week for 8 weeks. The exercises included mat and equipment-based exercises, focusing on core stabilization, breathing control, and postural alignment. Exercise difficulty was progressively increased throughout the intervention period.
  Interventions: Behavioral: Pilates
- Cervical Stabilization Exercise Group (Active Comparator): Participants in this group performed cervical stabilization exercises at home twice daily for 8 weeks.
  Interventions: Behavioral: Cervical stabilization exercise

INTERVENTIONS:
Behavioral: Pilates — Participants in this group performed Pilates exercises twice a week for 8 weeks. The exercises included mat and equipment-based exercises, focusing on core stabilization, breathing control, and postural alignment. Exercise difficulty was progressively increased throughout the intervention period.
  Arms: Pilates Exercise Group
Behavioral: Cervical stabilization exercise — Participants in this group performed cervical stabilization exercises at home twice daily for 8 weeks. The exercises included chin tucks, cervical extensions, shoulder elevations, and scapular retractions.
  Arms: Cervical Stabilization Exercise Group

SUMMARY:
This study aims to investigate and compare the effects of 8-week Pilates exercises and cervical stabilization exercises on pain, posture, range of motion, quality of life, and body composition in individuals with forward head posture (FHP). FHP is a common postural disorder characterized by the anterior displacement of the head relative to the cervical spine. This condition can lead to neck pain, muscle tension, and limited movement.

The study will include participants aged 18-50 years with FHP. Participants will be randomly assigned to one of two groups: the Pilates group or the cervical stabilization exercise group. The Pilates group will participate in Pilates exercises twice a week for 8 weeks under the supervision of a physiotherapist. The cervical stabilization exercise group will perform cervical stabilization exercises at home for the same duration.

The primary objective of this study is to compare the effects of Pilates and cervical stabilization exercises on FHP. Participants' posture, neck pain, range of motion, quality of life, and body composition will be measured before and after the 8-week intervention. These measurements will be used to evaluate and compare the effectiveness of the two exercise methods on FHP.

This study seeks to investigate the effectiveness of Pilates in the treatment of FHP and contribute to the scientific literature in this field. The findings may help determine the most appropriate exercise method for individuals with FHP.

DETAILED DESCRIPTION:
This study will be designed as an 8-week randomized controlled trial (RCT) to compare the effects of Pilates and cervical stabilization exercises (CSE) on forward head posture (FHP) in adult participants. Based on the understanding that proper posture is essential to maintain musculoskeletal balance and minimize excessive mechanical strain, the study will address the increasing prevalence of FHP-a problem exacerbated by sedentary lifestyles, prolonged screen use, and occupational demands. In FHP, the head is displaced forward relative to the cervical spine, disrupting the natural spinal curvature, which can lead to neck pain and altered muscle activation patterns.

The trial will be conducted in a controlled clinical setting at a physiotherapy center in Antalya, Turkey, in accordance with CONSORT 2010 guidelines. Robust randomization and blinded outcome assessments will be employed to ensure methodological rigor, and quality assurance protocols-such as regular equipment calibration and data audits-will be implemented to maintain data integrity.

Participants randomized to the Pilates intervention will participate in supervised sessions twice per week, each lasting 60 minutes, consisting of a 10-minute warm-up, a graduated main exercise phase, and a 10-minute cool-down. During the first four weeks, sessions will emphasize mat-based exercises focusing on core engagement, controlled breathing, and alignment. Beginning in Week 2, additional equipment (e.g., Pilates balls and 1-kg dumbbells) will be introduced, with resistance bands incorporated from Week 4 and further modified in Week 6 to progressively challenge participants. The control group will perform a daily CSE regimen (including chin tuck, cervical extension, shoulder elevation, and scapular retraction) structured into two sets designed to support neuromuscular control and postural stability. Both groups will receive ergonomic guidelines for daily posture management.

Data collection will be managed by trained physiotherapists who will adhere to strict protocols and perform regular device calibrations. Data analysis will be conducted using IBM SPSS Statistics (v29.0), employing appropriate statistical tests and calculating effect sizes, with a 95% confidence interval (p < 0.05) determining statistical significance. A comprehensive quality assurance plan-including regular audits, predefined data validation rules, and a maintained data dictionary-will further ensure the robustness and reliability of the findings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years.
* Craniovertebral angle (CVA) < 54°
* Sedentary lifestyle

Exclusion Criteria:

* History of spinal surgery (cervical/thoracic/lumbar) or neurological disorders.
* Acute or severe cervical trauma (e.g., fractures, whiplash injuries).
* Spinal deformities (e.g., scoliosis, kyphosis).
* Recent physiotherapy/manual therapy (within the past 6 months).
* Regular use of analgesics, muscle relaxants, or steroids.
* Active participation in regular exercise

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle (CVA) | Baseline (week 0) and after the 8-week intervention (week 8).
  The craniovertebral angle (CVA), a key metric and a widely used measure for assessing forward head posture (FHP), will be evaluated using standardized digital photogrammetry. Lateral photographs will be captured using a Fujifilm XT-3 mirrorless camera equipped with a 35mm lens. The CVA will be calculated as the angle between a line connecting the tragus and C7 markers and a horizontal reference line parallel to the floor. Higher CVA values will indicate a less severe forward head posture, reflecting better postural alignment.
Neck Pain Intensity | Baseline (week 0) and after the 8-week intervention (week 8).
  Neck pain intensity will be assessed using the Visual Analog Scale (VAS), a 10 cm line ranging from 0 (no pain) to 10 (unbearable/most severe pain). Participants will be instructed to rate their neck-specific discomfort on this scale. Lower scores will indicate less pain, while higher scores will indicate more severe pain.

SECONDARY OUTCOMES:
Posture | Baseline (week 0) and after the 8-week intervention (week 8)
  Posture will be assessed using the New York Posture Rating Scale (NYPRS). This method, also known as New York Posture Analysis Method (NYPAY), scores 13 body regions (head, neck, shoulders, back, waist, abdomen, pelvis, and feet) from posterior and lateral views. For each region, postural deviations will be scored observationally: 5 points for good posture, 3 points for moderately impaired posture, and 1 point for severely impaired posture. The body regions assessed include: head, neck, shoulders, back, waist, abdomen, pelvis, and feet. Total scores will be calculated by summing the scores across all 13 regions, resulting in a range from 13 (worst possible posture) to 65 (best possible posture). For interpretation, total NYPRS scores are categorized as follows: ≥45 points "very good", 40-44 points "good", 30-39 points "medium", 20-29 points "weak", and ≤19 points "bad" posture.. Therefore, higher total scores will indicate better overall posture.
Cervical Range of Motion (ROM) | Baseline (week 0) and after the 8-week intervention (week 8)
  Cervical range of motion (ROM), encompassing flexion, extension, lateral flexion, and rotation, will be measured using a standard universal goniometer. Maximum ROM angles will be recorded in degrees. For cervical ROM, higher values will indicate a greater range of motion, which is generally considered a better outcome.
SF-36 Quality of Life Questionnaire | Baseline (week 0) and after the 8-week intervention (week 8)
  Quality of life will be assessed using the Short Form-36 (SF-36) questionnairea comprehensive questionnaire evaluating different aspects of quality of life (physical, mental, social, etc.). This 36-item scale evaluates participants' health status over the past 4 weeks. The SF-36 includes eight subscales: physical functioning, role-physical, role-emotional, energy/vitality, mental health, social functioning, pain, and general health perceptions. Each subscale yields a score ranging from 0 to 100, where higher scores will indicate better quality of life in the respective domain.
Body Mass Index (BMI) | Baseline (week 0) and after the 8-week intervention (week 8)
  Body mass index (BMI) is a measure of body fat based on height and weight. It is calculated as weight in kilograms divided by height in meters squared (kg/m²). Weight will be measured using a calibrated digital scale, and height will be measured using a stadiometer.
Waist-to-hip ratio | Baseline (week 0) and after the 8-week intervention (week 8)
  The waist-to-hip ratio is calculated by dividing the waist circumference by the hip circumference (both measured in centimeters).
Waist circumference | Baseline (week 0) and after the 8-week intervention (week 8)
  Waist circumference is measured in centimeters at the level of the narrowest point between the lower rib and the iliac crest using a standard measuring tape. Three measurements will be taken at this point, and the average of these measurements will be recorded.
Hip circumference | Baseline (week 0) and after the 8-week intervention (week 8)
  Hip circumference is measured in centimeters at the level of the widest portion of the buttocks using a standard measuring tape. Three measurements will be taken at this point, and the average of these measurements will be recorded.
Chest circumference | Baseline (week 0) and after the 8-week intervention (week 8)
  Chest circumference is measured in centimeters at the level of the nipples using a standard measuring tape during normal breathing. Three measurements will be taken at this level, and the average of these measurements will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiolab Physiotherapy Center, Antalya, Alanya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All anonymized individual participant data (IPD) collected in this study, including demographic details, clinical measurements (CVA, pain scores, cervical ROM), SF-36 quality-of-life outcomes, and body composition data, will be shared upon reasonable request. Data will exclude raw imaging files, identifiable personal information, and non-anonymized records. Access requires submission of a scientifically valid proposal, a signed data access agreement, and compliance with ethical guidelines. Shared data will be deposited in a secure, open-access repository (e.g., Zenodo) with a DOI assigned for long-term availability. Data will remain accessible for at least 5 years post-publication. Requests will be reviewed by an independent committee to ensure alignment with research ethics and participant privacy protections (GDPR/Helsinki Declaration compliant).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD and supporting information will be available starting March 5, 2025 and will remain accessible for 5 years.
Access Criteria: Anonymized individual participant data (IPD) and supporting documents (study protocol, statistical analysis plan, informed consent form) will be provided upon request to researchers affiliated with academic institutions who have collaborated with the institution where the study was conducted and have signed a data use agreement. To access the data, researchers must submit their research proposals and request forms directly to yusufyasasin@gmail.com. The data will be stored on the secure server of the institution where the study was conducted. Access requests will be approved by the ethics committee of the institution where the study was conducted.